CLINICAL TRIAL: NCT00954681
Title: Open-Label Pilot Study of Quetiapine Treatment for Cannabis Dependence
Brief Title: Study of Quetiapine Treatment for Cannabis Dependence
Acronym: STUC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John Mariani MD, research psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5911; K23DA021209 (NIH)
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cannabis Dependence
Keywords: Cannabis; quetiapine
MeSH Terms: conditions — Marijuana Abuse | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- quetiapine treatment (Experimental): Open label treatment with quetiapine
  Interventions: Drug: quetiapine

INTERVENTIONS:
Drug: quetiapine — Quetiapine treatment from 25 mg daily to 300 mg twice daily
  Other Names: Seroquel

SUMMARY:
Marijuana is the most commonly used illicit drug in the United States. However, the treatment options for cannabis dependence are limited; notably, no effective pharmacotherapy has been developed. Conceptually, the ideal medication treatment for cannabis dependence would:

1. be safe when administered to patients actively using cannabis
2. reduce cannabis intake and promote abstinence
3. treat the symptoms of cannabis withdrawal
4. reduce craving and relapse risk
5. have a low abuse liability.

DETAILED DESCRIPTION:
Conceptually, the pharmacodynamic and clinical actions of quetiapine suggest that it may be useful for cannabis dependence. By antagonizing dopamine, quetiapine may interfere with the reinforcing effects of cannabis, while serotonin type 2A, histamine type 1, and adrenergic receptor antagonism may reduce cannabis withdrawal symptoms, primarily by sedating and anxiolytic effects. The proposed research project is an open-label pilot study to evaluate the tolerability and ideal target dosing range for quetiapine treatment of cannabis dependence over an eight-week period. The purpose of this pilot study is to obtain preliminary data regarding the potential efficacy, tolerability and safety of quetiapine treatment of cannabis dependence before conducting a larger double-blind trial.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-65
2. Meets DSM-IV criteria for current cannabis dependence
3. Seeking treatment for cannabis dependence
4. Reports using cannabis an average of five days per week over the past 28 days
5. Capable of giving informed consent and complying with study procedures

Exclusion Criteria:

1. Lifetime history of DSM-IV diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder
2. Current DSM-IV criteria for any other psychiatric disorder that may, according to the investigator's judgment, require either pharmacological or non-pharmacological intervention over the course of the study
3. Receiving prescribed psychotropic medication
4. Known history of allergy, intolerance, or hypersensitivity to quetiapine
5. Pregnancy, lactation, or failure to use adequate contraceptive methods in female patients who are currently engaging in sexual activity with men
6. Unstable medical conditions, such as poorly controlled diabetes or hypertension, which might make participation hazardous
7. Current DSM-IV diagnosis of substance dependence other than cannabis or nicotine dependence
8. Are legally mandated to participate in a substance use disorder treatment program
9. Increased risk for suicide
10. Diabetes (whether controlled or not), hyperglycemia (fasting glucose > 100 mg/dl), obesity (BMI > 30) and elevated lipids (cholesterol > 200 mg/dl; triglycerides > 150 mg/dl).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Mariani, MD, Principal Investigator — Columbia University
Locations (1):
- Substance Treatment Research Service (STARS) of Columbia University, New York, New York, United States

REFERENCES:
- See also: Substance Treatment Research Service (STARS) of Columbia University — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quetiapine Treatment
Started | 15
Completed | 10
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Quetiapine Treatment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 28.2 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 3
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Quetiapine
Description: Mean maximum tolerated dose of quetiapine
Time Frame: assesssed daily during 8 weeks of study, mean maximum tolerated dose reported
Population: Mean maximum dose of quetipaine achieved
Measure: Mean (Full Range); unit: milligrams
Groups:
- Open-Label Quetiapine Treatment: Participants receiving quetiapine under open-label conditions.
Arm/Group | Open-Label Quetiapine Treatment
Number analyzed (Participants) | 15
milligrams | 197 [25 to 600]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Quetiapine Treatment
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 12/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine Treatment (N=15)
fatigue (Nervous system disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No